CLINICAL TRIAL: NCT07170436
Title: Brain Areas of Cognitive Functions: a Study in Awake Surgery
Acronym: BRAIN-MAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/25/0226; ID-RCB (Other: 2025-A01307-42)
Record Dates: First submitted 2025-09-03; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Tumor
Keywords: surgery; awake surgery; brain; brain tumor; brain area
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pré-End (No Intervention): The day before surgery, brain tumor patients will be offered long-form cognitive tests. If the results of the cognitive tests are not consistent with the literature, this suggests that the tumor is affecting pre-contact time perception. These patients will not be tested during surgery.
- Pré-Per (Experimental): The day before surgery, brain tumor patients will be offered long-form cognitive tests. If the results of the cognitive tests are consistent with the literature, the short-form cognitive tests will be offered during awake surgery.
  Interventions: Behavioral: Short version of cognitive testing during surgery

INTERVENTIONS:
Behavioral: Short version of cognitive testing during surgery — Cognitive testing in 3 blocks of 3 minutes during awake surgery
  Arms: Pré-Per

SUMMARY:
This research project focuses on low-level cognitive functions such as perception (auditory, visual, etc.) and high-level cognitive functions (memory, language, temporal estimation, etc.). It aims to better understand the brain bases of these functions as well as their overlap (i.e., brain bases considered to be involved in different functions).

To this end, various cognitive tasks will be performed before and during awake brain surgery, allowing us to determine the involvement of different areas in the task being performed. Comparing performance between the pre-test and the intraoperative test will help determine the potential involvement of the tested area.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a brain tumor
* Aged 18 to 75 years
* Signed informed consent
* Vision that is corrected or adequate for the purposes of an experiment with visual stimuli
* Hearing that is corrected or adequate for the purposes of an experiment with auditory stimuli
* No known oculomotor disorder
* Person affiliated with or benefiting from a social security scheme.
* Free, informed, and written consent signed by the participant and the investigator (no later than the day of inclusion and before any examination required by the research)

Exclusion Criteria:

* Participants under protected status: guardianship, legal safeguard proceedings, or whose consent to participate in the experiment could be due to a severely altered psychological state, as determined by the medical team responsible for the surgery.
* History of neurological disease affecting the central nervous system (Parkinson's, Alzheimer's, history of stroke or cerebral infarction)
* Pregnant and/or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-11-08 (Estimated)

PRIMARY OUTCOMES:
development of an atlas mapping the brain regions involved in each major cognitive function | One day after the inclusion
  Analysis of the percentage of "yes" responses during the intraoperative phase, taking into account the expected probability based on preoperative results. Preoperative performance data allows to determine an expected performance level during the intraoperative phase.

SECONDARY OUTCOMES:
Number of tests | One day after the inclusion
  number of tests for which a brain area is considered to be involved during the analysis of the primary criterion for the pre-per group
Location of brain tumors | one day after the inclusion
  The MRI images of patients in the Pre-End group will be analyzed. It will be possible to determine whether their tumors overlap in a specific area, which could indicate that this area is essential for the process being studied.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neurochirurgie, Hôpital Pierre Paul Riquet, Place du Docteur Baylac, Toulouse, Oui, France

IPD SHARING:
Plan to Share IPD: No